CLINICAL TRIAL: NCT01611428
Title: A Single Dose, Open-label, Randomized Two-period Crossover Study in Healthy Young Subjects to Assess the Absolute Bioavailability of Ipragliflozin
Brief Title: Absolute Bioavailability Study With Ipragliflozin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Europe B.V. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 1941-CL-0057; 2010-023813-77 (EudraCT Number)
Record Dates: First submitted 2012-05-31; First posted 2012-06-05 (Estimated); Last update posted 2012-06-05 (Estimated); Status verified 2012-05

CONDITIONS: Bioavailability of Ipragliflozin; Healthy Subjects
Keywords: Ipragliflozin; Healthy; Absolute Bioavailability; Pharmacokinetics
MeSH Terms: interventions — ipragliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ipragliflozin - oral (Experimental): open label
  Interventions: Drug: Ipragliflozin
- Ipragliflozin - i.v. (Experimental): open label
  Interventions: Drug: Ipragliflozin

INTERVENTIONS:
Drug: Ipragliflozin — Oral and Intravenous (i.v.)
  Other Names: ASP1941

SUMMARY:
A study to assess the absolute bioavailability of ipragliflozin in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) more than or equal to 18.5 and less than 30.0 kg/m2

Exclusion Criteria:

* Any of the liver function tests above the upper limit of normal.
* Abnormal pulse and/or blood pressure measurements at the pre-study visit as follows: Pulse <40 or >90 bpm; mean systolic blood pressure >140 mmHg; mean diastolic blood pressure >90 mmHg (blood pressure measurements taken in triplicate after subject has been resting in supine position for 5 min; pulse will be measured automatically)
* A QTc interval of >430 ms (males) or > 450 ms (females) consistently after duplicate measurements, a history of unexplained syncope, cardiac arrest, unexplained cardiac arrhythmias or torsades de pointes, structural heart disease, or a family history of Long QT Syndrome (LQTS)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2011-06; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Assessment of the absolute bioavailability after a single oral dose of ipragliflozin | 6 days

SECONDARY OUTCOMES:
Evaluation of pharmacokinetics of ipragliflozin and its metabolite after a single oral dose and after an i.v. administration of ipragliflozin | 6 days
  AUClast (Area under the plasma concentration-time curve up to the last quantifiable sample), Cmax (Maximum plasma concentration), t1/2 (Apparent Terminal Elimination Half-life) and tmax (Time to Attain Cmax)
Evaluation of the safety and tolerability of a single oral dose of ipragliflozin assessed by recording adverse events, laboratory assessments, vital signs and electrocardiograms (ECGs) | 3 days
Evaluation of the safety and tolerability of an i.v. administration of ipragliflozin assessed by recording adverse events, laboratory assessments, vital signs and electrocardiograms (ECGs) | 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Study Manager, Study Director — Astellas Pharma Europe B.V.
Locations (1):
- Leeds, United Kingdom